CLINICAL TRIAL: NCT05297552
Title: An Open-label, Single-arm, Multi-center, Phase II Study to Evaluate the Efficacy and Safety of RC48-ADC Combined With JS001 in Perioperative Treatment of Muscle-Invasive Bladder Cancer
Brief Title: A Study of RC48-ADC Combined With JS001 For Perioperative Treatment of Muscle-Invasive Bladder Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C017
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Muscle Invasive Bladder Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC + JS001 (Experimental): Participants received 6 preoperative cycles of RC48-ADC PLUS JS001, followed by surgery, followed by up to 20 cycles of postoperative JS001.
  Interventions: Drug: RC48-ADC; Drug: JS001

INTERVENTIONS:
Drug: RC48-ADC — Drug: RC48-ADC 2.0 mg/kg by intravenous (IV) infusion, given on Day 1 of each 14-day cycle
Drug: JS001 — Drug: JS001 3.0 mg/kg by intravenous (IV) infusion, given on Day 1 of each 14-day cycle

SUMMARY:
This study will evaluate the efficacy and safety of intravenous RC48-ADC combined with JS001 in perioperative treatment of muscle-invasive bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Male or female, Age ≥ 18 years.
* Predicted survival ≥ 12 weeks.
* Histologically confirmed diagnosis of muscle invasive bladder cancer (MIBC) .Naive of antitumor systematic treatment or radiotherapy.
* Have clinically non-metastatic bladder cancer (cT2-T4a, N0-1, M0) determined by imaging.
* Be deemed eligible for Radical Cystectomy (RC) + Pelvic Lymph Node Dissection (PLND).
* HER2 expressing (i.e. IHC 1+ 2+ or 3+) as confirmed by the local lab.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Adequate organ function, evidenced by the following laboratory results within 7 days prior to the study treatment.
* Male and female participants are eligible to participate if they agree to the contraception use as per study protocol.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Has received other antitumor therapy before planned start of trial treatment.
* History of major surgery within 4 weeks of planned start of trial treatment.
* Diagnosed with HBsAg, HBcAb positive and HBV DNA copy positive, or HCVAb positive, or HIVAb positive.
* Has received a live virus vaccine within 4 weeks of planned start of trial treatment.
* NYHA Class III heart failure.
* Suffering from active infection requiring systemic treatment.
* Uncontrolled hypertension, diabetes, Interstitial lung Disease, or COPD;
* Treated with systemic treatment (e.g. immunomodulators, corticosteroids or immunosuppressants) for the autoimmune disease within 2 years prior to the study treatment.
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or cancers with a similar curative outcome as those mentioned above.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Pregnancy or lactation.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | Up to approximately 16 Weeks (Time of surgery)
  pCR rate is defined as the percentage of participants having pCR. pCR is defined as absence of viable tumor (pT0pT0N0) in examined tissue from RC and PLND.

SECONDARY OUTCOMES:
Rate of Pathologic Response | Up to approximately 16 Weeks (Time of surgery)
  No residual tumor (ypT0N0) and partial response (ypTis-1N0) in surgical specimen.
1-year Disease Free Survival Rate | From approximately 16 Weeks up to approximately 12 Months.
  The percentage of participants disease free on 1 year after surgery.
Objective Response Rate (ORR) | Up to approximately 12 Weeks.
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)
Overall Survival (OS) | Up to approximately 60 Months.
  Overall survival is defined as the time from enrollment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Ph.D, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided